CLINICAL TRIAL: NCT02863601
Title: Impact of Pregnancy on Buprenorphine Pharmacokinetics and Pharmacodynamics
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steve N. Caritis, MD, Professor, University of Pittsburgh
Other Study IDs: PRO15120442; STUDY19030255 (Other: PittPRO)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Opiate Addiction; Pregnancy
Keywords: Buprenorphine; Opiate Substitution Treatment
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous Blood, Hair, Urine, Saliva, Placenta, Umbilical Cord Blood/Tissue, Postpartum Breast Milk
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pregnant: pregnant women prescribed buprenorphine
- postpartum: Postpartum women prescribed buprenorphine

SUMMARY:
The primary purpose of this study is to determine whether buprenorphine and metabolite exposure (reflected as the dose-adjusted plasma concentration x time curve [AUC]) differs during pregnancy and between pregnancy and the postpartum state.The study will define the pharmacokinetics of buprenorphine and determine if there is a better way to gauge dosing based on objective, physiological parameters of satiety. The study will define neonatal exposure to buprenorphine through breast milk.

DETAILED DESCRIPTION:
Currently, the standard of care for an opioid-dependent pregnant woman in most institutions is methadone, however, buprenorphine (BUP) is also used for this indication, as it is FDA-approved for opioid addiction although not specifically for pregnant women. There has been increasing evidence that BUP may have comparable efficacy to methadone, and may have fewer severe neonatal complications especially neonatal abstinence syndrome (NAS) and decreased severity of adverse reactions. The dosing of BUP currently is based on studies in men and non-pregnant women (adjusted to the patient's symptomatology using the Clinical Opiate Withdrawal (COW) score, some of which is subjective and some based on objective physiological parameters) and limited animal data that related plasma concentrations of BUP to the degree of saturation of the µ receptor in the brain.

The study team will define the pharmacokinetics and limited pharmacodynamics of BUP in early and late pregnancy and the postpartum period and determine what contributes to the variation in plasma concentrations and response and will also relate plasma concentrations of BUP and its major metabolites to physiologic parameters that can be used to gauge the amount of drug in mother's plasma. It is expected to demonstrate that higher doses of BUP are needed throughout pregnancy and that the dosing regimen can be adjusted using patient covariates and biophysical measurements in addition to the COW scores.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 45 years
* Currently on a stable two, three, four, or five times daily dose of sublingual BUP
* Willingness to participate in at least one pharmacokinetic(PK)/pharmacodynamics study either during pregnancy or in postpartum*
* Gestational age < 19 6/7 weeks *
* Singleton gestation
* Able to give informed consent and undergo study procedures
* Willing to have urine samples screened for the presence of alcohol, barbiturates, opiates, cocaine (or metabolites), benzodiazepines, synthetic opioids and phencyclidine

  * Requirement applies only to those subjects in the PK study

Exclusion Criteria:

* Major fetal anomalies or malformations
* HIV or AIDS
* Comorbid dependence on benzodiazepines or other central nervous system depressants (including anti-seizure medications)
* Taking medication known to interfere with buprenorphine metabolism
* Active or chronic suicidal or homicidal ideation or attempts
* Elevated liver enzymes (AST, alanine aminotransferase (ALT) > 2 times normal) *
* Creatinine > 1.5 mg/dl *
* Delivery at other institution where outcome data or samples cannot be obtained on mother and baby
* Active use of non- prescribed opiates/opioids detected during the urine drug screen performed within 1 week prior to each PK visit *
* Hematocrit <28 *

  * Requirement applies only to those subjects in the PK study

There are several parts to this study and subjects may participate in the PK study and/or one or more procedures other than the PK study. All parts of the study (Parts A-E) are described in the attached protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample of pregnant women who are receiving sublingual BUP (subutex) in a supervised hospital or outpatient clinical setting because of their opiate addiction.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Exposure to BUP (AUC) during pregnancy and the post-partum state | Between 8 weeks 0/7 days and 20 weeks 6/7 days gestational age; between 21 weeks 0/7 days and 35 weeks 6/7 days gestational age; 4-6 weeks postpartum
  We will define the pharmacokinetics of BUP in early and late pregnancy and the postpartum period and determine what contributes to the variation in plasma concentrations and response.

CONTACTS AND LOCATIONS:
Overall Officials: Steve N Caritis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Donna DeAngelis, Pittsburgh, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT02863601/Prot_SAP_020.pdf